CLINICAL TRIAL: NCT02489188
Title: Gait Asymmetry in Orthopaedic Conditions of the Lower Extremity Assessed Using Portable and Laboratory Based Systems: Cross-sectional Observational Single-centre Pilot Study
Brief Title: Gait Asymmetry Assessed Using Portable Gait Analysis System
Acronym: Asymmetry
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-139
Record Dates: First submitted 2015-06-23; First posted 2015-07-02 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Ankle Osteoarthritis; Knee Osteoarthritis; Hip Osteoarthritis; Lumbar Spine Stenosis; Muscle Contracture
Keywords: gait asymmetry; joint angles
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Contracture | interventions — Arthroplasty; Musculoskeletal Manipulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- ankle osteoarthritis: patients with ankle osteoarthritis scheduled for arthroplasty
  Interventions: Procedure: arthroplasty; Other: manual therapy
- knee osteoarthritis: patients with knee osteoarthritis scheduled for arthroplasty
  Interventions: Procedure: arthroplasty; Other: manual therapy
- hip osteoarthritis: patients with hip osteoarthritis scheduled for arthroplasty
  Interventions: Procedure: arthroplasty; Other: manual therapy
- lumbar spinal stenosis: patients with lumbar spinal stenosis scheduled for lumbar spinal stenosis decompression
  Interventions: Other: manual therapy; Procedure: lumbar spinal stenosis decompression
- muscle contracture: patients with functionally limited range of motion at the knee because of muscle contracture scheduled for manual therapy
  Interventions: Other: manual therapy
- healthy subjects: healthy subjects

INTERVENTIONS:
Procedure: arthroplasty — patients, who are scheduled for arthroplasty, will be measured before and on average 6 months after surgery
  Groups: ankle osteoarthritis; hip osteoarthritis; knee osteoarthritis
Other: manual therapy — patients, who are scheduled for manual therapy, will be measured before, immediately and on average 1 week after treatment
  Groups: ankle osteoarthritis; hip osteoarthritis; knee osteoarthritis; lumbar spinal stenosis; muscle contracture
Procedure: lumbar spinal stenosis decompression — patients, who are scheduled for lumbar spinal stenosis decompression, will be measured before and on average 6 months after surgery
  Groups: lumbar spinal stenosis

SUMMARY:
To date, detailed analysis of movement patterns in orthopaedic conditions are mainly performed in research projects. Because these tests are time consuming, they are not feasible in clinical routine or in standard examinations. Novel technologies allow capturing detailed movement patters within a few minutes. The aim of this regional study is to compare aspects of movement tasks measured using a mobile gait analysis system to those measured using laboratory based systems and to determine aspects of gait patterns relevant for different orthopaedic conditions. Moreover, the researchers will investigate if these relevant aspects can be altered using surgical treatment or manual therapy.

DETAILED DESCRIPTION:
This is a cross-sectional study. Pre- and post-treatment data will only be collected in patients undergoing routine orthopaedic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years, for patients: diagnosed osteoarthritis at the ankle, knee or hip, lumbar spinal stenosis or limited range of motion at the knee

Exclusion Criteria:

* Body mass index > 35kg/m2
* Use of walking aids
* Inability to walk for 6 minutes
* Neuromuscular disorders affecting gait
* Cardiovascular disease
* Inability to follow procedures due to psychological disorders or dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients visiting the outpatient clinic or are scheduled for arthroplasty or LSS decompression at the University Hospital Basel and from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
symmetry index | up to 6 months
  gait asymmetry assessed using a portable and laboratory gait analysis systems

SECONDARY OUTCOMES:
change in symmetry index | up to 6 months
  changes in gait asymmetry assessed using a portable and laboratory gait analysis systems
maximum isokinetic joint moment [Nm] | up to 6 months
  isokinetic muscle strength
relative electromyographic (EMG) intensity | up to 6 months
  electromyographic activity normalised to activity during maximum voluntary contraction
differences between maximum flexion and extension [degrees] | up to 6 months
  passive range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Horstmann T, Listringhaus R, Haase GB, Grau S, Mundermann A. Changes in gait patterns and muscle activity following total hip arthroplasty: a six-month follow-up. Clin Biomech (Bristol). 2013 Aug;28(7):762-9. doi: 10.1016/j.clinbiomech.2013.07.001. Epub 2013 Jul 29. PMID 23906936
- [Background] Horstmann T, Listringhaus R, Brauner T, Grau S, Mundermann A. Minimizing preoperative and postoperative limping in patients after total hip arthroplasty: relevance of hip muscle strength and endurance. Am J Phys Med Rehabil. 2013 Dec;92(12):1060-9. doi: 10.1097/PHM.0b013e3182970fc4. PMID 23739275
- [Background] Horstmann T, Vornholt-Koch S, Brauner T, Grau S, Mundermann A. Impact of total hip arthroplasty on pain, walking ability, and cardiovascular fitness. J Orthop Res. 2012 Dec;30(12):2025-30. doi: 10.1002/jor.22163. Epub 2012 May 31. PMID 22653634
- [Background] Mundermann A, Mundermann L, Andriacchi TP. Amplitude and phasing of trunk motion is critical for the efficacy of gait training aimed at reducing ambulatory loads at the knee. J Biomech Eng. 2012 Jan;134(1):011010. doi: 10.1115/1.4005540. PMID 22482665
- [Background] Mundermann A, Asay JL, Mundermann L, Andriacchi TP. Implications of increased medio-lateral trunk sway for ambulatory mechanics. J Biomech. 2008;41(1):165-70. doi: 10.1016/j.jbiomech.2007.07.001. Epub 2007 Aug 3. PMID 17678933
- [Background] Fisher DS, Dyrby CO, Mundermann A, Morag E, Andriacchi TP. In healthy subjects without knee osteoarthritis, the peak knee adduction moment influences the acute effect of shoe interventions designed to reduce medial compartment knee load. J Orthop Res. 2007 Apr;25(4):540-6. doi: 10.1002/jor.20157. PMID 17205556
- [Background] Mundermann A, Dyrby CO, Andriacchi TP. Secondary gait changes in patients with medial compartment knee osteoarthritis: increased load at the ankle, knee, and hip during walking. Arthritis Rheum. 2005 Sep;52(9):2835-44. doi: 10.1002/art.21262. PMID 16145666
- [Background] Mundermann A, Dyrby CO, Hurwitz DE, Sharma L, Andriacchi TP. Potential strategies to reduce medial compartment loading in patients with knee osteoarthritis of varying severity: reduced walking speed. Arthritis Rheum. 2004 Apr;50(4):1172-8. doi: 10.1002/art.20132. PMID 15077299
- [Background] Nuesch C, Huber C, Paul J, Henninger HB, Pagenstert G, Valderrabano V, Barg A. Mid- to Long-term Clinical Outcome and Gait Biomechanics After Realignment Surgery in Asymmetric Ankle Osteoarthritis. Foot Ankle Int. 2015 Aug;36(8):908-18. doi: 10.1177/1071100715577371. Epub 2015 Mar 20. PMID 25795650
- [Background] Nuesch C, Valderrabano V, Huber C, Pagenstert G. Effects of supramalleolar osteotomies for ankle osteoarthritis on foot kinematics and lower leg muscle activation during walking. Clin Biomech (Bristol). 2014 Mar;29(3):257-64. doi: 10.1016/j.clinbiomech.2013.12.015. Epub 2013 Dec 31. PMID 24445126
- [Background] Nuesch C, Barg A, Pagenstert GI, Valderrabano V. Biomechanics of asymmetric ankle osteoarthritis and its joint-preserving surgery. Foot Ankle Clin. 2013 Sep;18(3):427-36. doi: 10.1016/j.fcl.2013.06.002. Epub 2013 Jul 24. PMID 24008209
- [Background] Nuesch C, Valderrabano V, Huber C, von Tscharner V, Pagenstert G. Gait patterns of asymmetric ankle osteoarthritis patients. Clin Biomech (Bristol). 2012 Jul;27(6):613-8. doi: 10.1016/j.clinbiomech.2011.12.016. Epub 2012 Jan 18. PMID 22261013